CLINICAL TRIAL: NCT00268411
Title: Phase II Randomisee Dans Les Adenocarcinomes Metastatiques Du Pancreas: Gemox Et Gemox Simplifie. [GEMOX]
Brief Title: Gemcitabine and Oxaliplatin in Treating Patients With Metastatic Pancreatic Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000453849; GERCOR-D04-1-GEMOX; EU-20569; SANOFI-GERCOR-D04-1-GEMOX
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2008-05-27 (Estimated); Status verified 2007-05

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Oxaliplatin

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. It is not yet known whether giving both of these drugs on the same day is more effective than giving them on different days.

PURPOSE: This randomized phase III trial is studying two different schedules of gemcitabine and oxaliplatin to compare how well they work in treating patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the objective response rate in patients with metastatic adenocarcinoma of the pancreas treated with two different schedules of gemcitabine hydrochloride and oxaliplatin.

Secondary

* Compare the clinical benefits and tolerability of these regimens in these patients.
* Compare the progression-free and overall survival of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to the participating center and ECOG performance status (0 or 1 vs 2). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive gemcitabine hydrochloride IV over 100 minutes on day 1 and oxaliplatin IV over 2 hours on day 2.
* Arm II: Patients receive gemcitabine hydrochloride IV over 100 minutes followed by oxaliplatin IV over 2 hours on day 1.

In both arms, treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 80 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the pancreas

  * Metastatic disease
* Measurable disease (primary tumor or metastasis)

  * At least 1 cm in diameter by spiral CT scan
* No ampulla of Vater carcinoma or biliary adenocarcinoma
* No known brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 or Karnofsky PS 60-100%
* Life expectancy more than 12 weeks
* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Alkaline phosphatase < 5 times normal
* Bilirubin < 1.5 times normal
* Creatinine < 1.5 times normal
* No pre-existing neuropathy
* No unstable or uncontrolled pain
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No serious cardiovascular disease
* No serious respiratory disease
* No uncontrolled or persistent hypercalcemia
* No psychological, familial, social, or geographical condition that would preclude study treatment
* No other active malignancy

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy
* No concurrent corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2004-09

PRIMARY OUTCOMES:
Objective response rate

SECONDARY OUTCOMES:
Clinical benefits and tolerability
Progression-free and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Louvet, MD, PhD, Study Chair — Hopital Saint Antoine
Locations (15):
- France (15):
  - Hopital Duffaut, Avignon
  - C.H.G. Beauvais, Beauvais
  - Hopital Drevon, Dijon
  - Centre Hospitalier de Dreux, Dreux
  - Centre Hospitalier Departemental, La Roche-sur-Yon
  - Hopital Saint - Louis, La Rochelle
  - Hopital Louis Pasteur - Le Coudray, Le Coudray
  - Clinique Victor Hugo, Le Mans
  - Polyclinique des Quatre Pavillons, Lormont
  - Clinique Saint Jean, Lyon
  - Hopital Saint Antoine, Paris
  - Hopital Tenon, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Polyclinique De Courlancy, Reims
  - C.H. Senlis, Senlis